CLINICAL TRIAL: NCT01697371
Title: Phase I-II Trial of Stereotactic Body Proton Therapy for Patients With Liver Metastases
Brief Title: Proton Therapy in the Treatment of Liver Metastases
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5120022
Record Dates: First submitted 2012-09-07; First posted 2012-10-02 (Estimated); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Liver Metastases
MeSH Terms: interventions — Protons; Proton Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Proton Radiation (Experimental)
  Interventions: Radiation: Proton; Radiation: Proton Radiation

INTERVENTIONS:
Radiation: Proton — All patients will receive 3 fractions in no more than 14 days at the following levels: Level I = 12 Gy per fraction, total dose=36 Gy.
  Level II = 16 Gy per fraction, total dose 48 Gy. Level III = 20 Gy per fraction, total dose 60 Gy. The dose per fraction to the PTV will start at dose level I (12 Gy), but may vary from 12 Gy to 20 Gy in 3 fractions over 14 days in 4 Gy increments
Radiation: Proton Radiation

SUMMARY:
Local control of hepatic metastases appears to be a major determinant of overall survival. However, many patients are not suitable for resection due to medical or surgical reasons. Therefore, there is an important role for a treatment that can provide the equivalent of tumor resection with minimal morbidity. Stereotactic body radiotherapy (SBRT) delivers an ablative regimen of highly focused external beam radiotherapy that targets one or more discrete extracranial lesions. Published reports using SBRT to treat liver metastases have shown actuarial local control rates ranging from 50-100% with higher doses associated with better local control.

In patients with metastatic liver disease, aggressive local therapy using modern radiotherapy techniques are promising and project to have a substantial role in the treatment of metastatic liver cancer to treat unresectable disease. The dosimetric advantage of proton therapy may lead to improved clinical outcomes with less morbidity, however, there is no clinical data to confirm this assertion. We thus propose a phase I study to determine the feasibility and safety of stereotactic body proton therapy in patients with liver metastases followed by a phase II study to determine the efficacy of such treatment on local control.

ELIGIBILITY:
Inclusion Criteria:

Pathologically confirmed non-lymphoma liver metastases or

New radiographic liver lesions consistent with metastases in patients with known pathologically confirmed non-lymphoma cancer

1-3 liver lesions measurable on CT/MRI or PET/CT performed within 6 weeks prior to study entry

Liver metastases measuring <5cm

Life expectancy >6 months

Disease outside the liver is allowed

Age ≥ 18

ECOG Performance Scale = 0-1

Adequate bone marrow function, defined as follows:

* Absolute neutrophil count (ANC) ≥ 1,000 cells/mm3 based upon CBC/differential obtained within 4 weeks prior to registration on study
* Platelets ≥ 60,000 cell/mm3 based upon CBC/differential obtained within 4 weeks prior to registration on study
* Hemoglobin ≥ 8.0 g/dl based upon CBC/differential obtained within 4 weeks prior to registration on study (Note: the use of transfusion or other intervention to achieve Hgb ≥ 8.0 is acceptable.)

Adequate kidney function (serum creatinine <2mg/dL) based on chemistry panel obtained within 4 weeks prior to registration on study

Adequate liver function, defined as total bilirubin <5 mg/dL, serum albumin >2.0g/dL, serum levels of liver enzymes < 5 times the upper limit of normal, and INR < 1.5

Previous liver resection or ablative therapy is permitted

Chemotherapy and/or targeted agent therapy must be completed at least 2 weeks prior to radiation and started at least 14 days after completion of SBPT Women of childbearing potential and male participants must practice adequate contraception

Patient must sign study specific informed consent prior to study entry

Pretreatment evaluations required for eligibility include:

* A complete history and general physical examination
* For women of childbearing potential, a serum or urine pregnancy test must be performed within 72 hours prior to registration
* INR, total bilirubin, albumin, alkaline phosphatase, ALT, AST within 4 weeks prior to study entry

Exclusion Criteria:

Prior invasive malignancy other than liver met primary (except non-melanomatous skin cancer) unless disease free for > 3years

Prior radiotherapy that would results in overlap of radiation fields

Prior radiotherapy to the liver

Severe, active co-morbidity that may impact survival

CNS metastases

Tense ascites requiring frequent paracentesis

Active liver infection

Pregnancy, nursing women, or women of child bearing potential, and men who are sexually active and not willing/able to use medically acceptable forms of contraception

Metastases location within 2cm of GI tract

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2012-08-22 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2033-09 (Estimated)

PRIMARY OUTCOMES:
Phase I of study: Number of participants with adverse events as a measure of safety and tolerability | The major analysis for reporting the initial results of treatment will be undertaken when each patient has been potentially followed for a minimum of 3 months

SECONDARY OUTCOMES:
Phase II -local control within irradiated fields at 2 years | The major analysis for reporting the initial results of treatment will be undertaken when each patient has been potentially followed for a minimum of 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Gary Yang, MD, Principal Investigator — gyang@llu.edu
Locations (1):
- Loma Linda University Medical Center, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kang JI, Sufficool DC, Hsueh CT, Wroe AJ, Patyal B, Reeves ME, Slater JD, Yang GY. A phase I trial of Proton stereotactic body radiation therapy for liver metastases. J Gastrointest Oncol. 2019 Feb;10(1):112-117. doi: 10.21037/jgo.2018.08.17. PMID 30788166